CLINICAL TRIAL: NCT03759457
Title: High Flow Nasal Cannula (HFNC) in COPD Patients With Persistent Hypercapnia After an Acute Exacerbation
Brief Title: High Flow Nasal Cannula and Hypercapnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief of the Respiratory nad Critical Care Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Iperpneumo
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Flow Nasal Cannula (Experimental): High Flow Nasal Cannula is a relatively new technique able to deliver both oxygen and high flow in order to improve oxygenation and waking out CO2 from the upper airways
  Interventions: Device: High Flow Nasal Cannula (AIRVO2)

INTERVENTIONS:
Device: High Flow Nasal Cannula (AIRVO2) — High-flow nasal cannula (HFNC) delivers oxygen flows of up to 60 L/min. The gas source (air/oxygen blender, ventilator, or turbine flow-generator) is connected via an active heated humidifier to a nasal cannula and allows FiO2 adjustment independently from the flow

SUMMARY:
In the present investigation, in 50 COPD with persistent hypercapnia after an acute exacerbation, the investigators want to assess the acceptability of HFNC and its effectiveness in further reducing the level of PaCO2, and to eventually verify the hypothesis, based on previous physiological studies, that the response to HFNC is dependent on the level of baseline hypercapnia and eventually on the presence of overlap syndrome. This latter parameters to eventually calculate the sample size and the target population to perform future definitive randomized long term trials vs NIV.

DETAILED DESCRIPTION:
Fifthy COPD patients inpatients recovering from an acute exacerbation of their disease and persisting hypercapnia, despite having reached a stabilization in pH (i.e. pH>7,35 and PaCO2>45 mmHg on 3 consecutive measurements) will be enrolled in the study after having signed a written informed consent OSA/COPD overlap syndrome was not considered and exclusion criteria and is defined as the presence of 15 or more obstructive respiratory events per hour of sleep, when a previous full night polysomnography (PSG) was available or from a positive Epworth questionnaire and a Body Mass Index>25 Cardiac decompensation, restrictive thoracic disorders, renal insufficiency, cancer, and neurological disease were considered exclusion criteria.

On day the patients will undergo a preliminary trial with HFNC to set the optimal flow, using the AIRVO2 (Fisher & Paykel Healthcare, Auckland, New Zealand). To this aim the patients will be asked to breathe keeping their mouth closed, as much as they could, at different levels of flow, starting from 20 L/min up to 40 if tolerated for a minimum of 15 minutes for each trial. At the end of this test the maximum level tolerated will be chosen as the flow to be set for the experimental procedure. Temperature will be set according to the patient's tolerance starting from 34C, up to 37C, while FiO2 will be kept constant to maintain an SaO2 between 92 and 94%.

From 9 am of day 2 to 9 am of day 5 (72 hours period), the patients will undergo HFNC for at least 8 hours/day and during the nightime. The nurse on shift will be in charge of supervising the adherence to this schedule and to report any violation of the protocol on a dedicated sheet. Every morning at 10 am (1 hour after HFNC suspension) Arterial Blood Gases (ABGs), effective hours of HFT and tolerance to the treatment as reported by the patient, using a dedicated scale where: )1. Very bad 2. Bad 3. Moderate 4. Good 5.very good) will be recorded

ELIGIBILITY:
Inclusion Criteria:

* inpatients recovering from an acute exacerbation of their disease
* persisting hypercapnia, despite having reached a stabilization in pH (i.e. pH>7,35 and PaCO2>45 mmHg on 3 consecutive measurements)

Exclusion Criteria:

* Cardiac decompensation,
* restrictive thoracic disorders,
* renal insufficiency,
* cancer,
* neurological disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-01-29 (Estimated); Study Completion 2019-01-29 (Estimated)

PRIMARY OUTCOMES:
changes in Arterial Blood Gases (ABGs) | immediately after intervention
  Arterial Blood Gases, namely arterial oxygen (PaO2) and carbon dioxyde (PaCO2) tension will be analyzed from a sample taken from the arterial artery

SECONDARY OUTCOMES:
tolerance to the treatment | immediately after intervention
  this will be assessed using a standardized 4 points scale where tolerance to the treatment as reported by the patient, where categorized as: )1. Very bad 2. Bad 3. Moderate 4. Good 5.very good

CONTACTS AND LOCATIONS:
Overall Officials: stefano nava, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Sant'Orsola Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
cannot release data prior to the termination of the study

REFERENCES:
- [Derived] Pisani L, Betti S, Biglia C, Fasano L, Catalanotti V, Prediletto I, Comellini V, Bacchi-Reggiani L, Fers SN. Effects of high-flow nasal cannula in patients with persistent hypercapnia after an acute COPD exacerbation: a prospective pilot study. BMC Pulm Med. 2020 Jan 13;20(1):12. doi: 10.1186/s12890-020-1048-7. PMID 31931776